CLINICAL TRIAL: NCT06634056
Title: Pneumonitis Prevention Protocol Using Pentoxifylline and α-tocopherol in Stage III Non-Small Cell Lung Cancer Patients Undergoing Chemoradiation
Acronym: P4-PACIFIC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 24-5340
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Non-Small Cell Lung Cancer; Radiation Induced Lung Injury (RILI)
Keywords: P4-PACIFIC; Radiation Induced Lung Injury (RILI); Non-Small Cell Lung Cancer; Pentoxifylline; α-Tocopherol (Vitamin E)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pentoxifylline; alpha-Tocopherol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Placebo Comparator): Participants in the control arm will start one placebo orally three times a day and another placebo orally two times a day on day one of radiotherapy and continue treatment for 6 months.
  Interventions: Other: Placebo
- Experimental Arm (Experimental): Participants in the experimental arm will start Pentoxifylline 400 mg orally three times a day and α-Tocopherol 400 IU orally two times a day on day one of radiotherapy and continue treatment for 6 months.
  Interventions: Drug: Pentoxifylline; Other: α-Tocopherol

INTERVENTIONS:
Drug: Pentoxifylline — Pentoxifylline 400 mg orally three times a day and α-Tocopherol IU orally two times a day on day one of radiotherapy and continue treatment for 6 months.
  Arms: Experimental Arm
Other: Placebo — One placebo orally three times a day and another placebo orally two times a day on day one of radiotherapy and continue treatment for 6 months.
  Arms: Control Arm
Other: α-Tocopherol — Pentoxifylline 400 mg orally three times a day and α-Tocopherol IU orally two times a day on day one of radiotherapy and continue treatment for 6 months.
  Arms: Experimental Arm

SUMMARY:
Currently, the standard of care treatment for newly diagnosed, inoperable stage III non-small cell lung cancer is radiotherapy (RT) with concurrent chemotherapy, followed by immune checkpoint inhibitors (ICI). RT is a highly effect local treatment. However, high doses of radiation used in curative settings can cause adverse side effects. The most common RT side effect in lung cancer is Radiation Induced Lung Injury (RILI), which can manifest as pneumonitis and/or pulmonary fibrosis. Lung injury can negatively impact patients' well-being and quality of life, and may lead to increased mortality. Risk of lung injury is particularly increased when patients are treated with a combination of treatments (i.e., RT, chemotherapy, and ICI). The drug Pentoxifylline (in combination with α-Tocopherol (Vitamin E)) has been shown to prevent/alter the progression of lung injury and there is a growing body of evidence to support the safety and efficacy of phosphodiesterase inhibitors in cancer treatment. The proposed study aims to determine if the addition of Pentoxifylline, given in combination with α-Tocopherol (Vitamin E), to standard of care treatment will reduce side effects related to lung injury and improve quality of life in this study population.

DETAILED DESCRIPTION:
This is a multi-centre, Phase II, double-blind, placebo-controlled randomized trial. Eligible participants will include newly diagnosed, inoperable Stage III patients with NSCLC who will be treated with radical intent concurrent chemoradiation therapy with planned consolidation immune checkpoint inhibitor (ICI) as per standard of care. Participants will be randomized in a 1:1 ratio between control arm (Placebos for 6 months) (Arm 1) and the experimental arm (Pentoxifylline/α-Tocopherol for 6 months) (Arm 2).

ELIGIBILITY:
Inclusion Criteria:

* Female and/or male aged ≥ 18 years.
* Histologically confirmed diagnosis of stage III NSCLC, planned for treatment with concurrent chemoradiation and consolidation immune checkpoint inhibitor as per standard of care with no medical contraindications to therapy.
* Patients with ECOG performance status 0-2 within 4 weeks of randomization.
* Adequate liver function (no evidence of Child-Pugh class C disease or cirrhosis) as per blood work done within 30 days of registration.
* Adequate kidney function (Creatinine clearance > 50 mL/min) as per blood work done within 30 days of registration.

Exclusion Criteria:

* Participation in another clinical study with an investigational product during the last 6 months prior to registration.
* Patients who will have surgery as part of curative treatment.
* Previous radiotherapy to intended treatment volumes in the thorax.
* Active pregnancy.
* Life expectancy of less than 12 months.
* Hypersensitivity to Pentoxifylline or other xanthines such as caffeine, theophylline and theobromine or tocopherol (vitamin E).
* Participant has a history of acute (within 3 months) myocardial infarction, coronary artery disease, or cardiac arrhythmias.
* Ongoing hemorrhage or major bleeding risk. Patients on antiplatelets agents and anticoagulants (Aspirin, Clopidogrel, Ticlopidine, Cilostazol, Dipyridamole, Heparin, Dalteparin, Enoxaparin and Warfarin) can be enrolled, but major bleeding events will be captured. Patients on Warfarin will need frequent monitoring of their coagulation time to adjust Warfarin dosage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-05-30 (Estimated); Primary Completion 2031-11-30 (Estimated); Study Completion 2032-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in risk of Lung Injury | 1 year
  To evaluate whether the addition of Pentoxifylline and α-Tocopherol changes the risk of lung injury within 12 months post radiotherapy. Lung injury as defined by Grade2+ pneumonitis.

SECONDARY OUTCOMES:
Change in Oncological Outcomes | 1 year
  To evaluate whether the addition of Pentoxifylline and α-Tocopherol changes oncological outcomes of progression free survival and overall survival. Progression free survival as measured by RECIST 1.1.
Change in Grade 3-5 treatment related toxicities | 1 year
  To evaluate whether the addition of Pentoxifylline and α-Tocopherol changes the incidence of Grade 3-5 treatment (chemoRT + ICI) related toxicity. Grade 3-5 treatment related toxicity measured as per CTCAE version 5.0.
Change in Quality of Life | 1 year
  To evaluate whether the addition of Pentoxifylline and α-Tocopherol changes quality of life, as measured by FACT-LCS (version 4) scores

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network - Princess Margaret Cancer Centre, Toronto, Ontario, Canada